CLINICAL TRIAL: NCT00049725
Title: A Study of Daclizumab in Chronic Immune Thrombocytopenia (ITP)
Brief Title: Daclizumab to Treat Chronic Immune Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030046; 03-CC-0046
Record Dates: First submitted 2002-11-12; First posted 2002-11-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-12

CONDITIONS: Thrombocytopenia
Keywords: Autoimmune Disease; Monoclonal Antibody Therapy; Anti-IL2 Receptor; Platelets; Monoclonal Antibody; Immune Thrombocytopenia; ITP
MeSH Terms: conditions — Thrombocytopenia; Autoimmune Diseases; Purpura, Thrombocytopenic, Idiopathic | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This study will evaluate the effectiveness of the drug daclizumab for treating patients with chronic immune thrombocytopenia (ITP), a disease in which the immune system destroys platelets (blood cells involved in the clotting process). Patients with ITP have abnormal bruising and bleeding; severe disease can be life-threatening. For many patients, standard drug treatments are not effective, and many of the drugs used may have significant side effects with long-term use. Daclizumab is a genetically engineered antibody that suppresses the immune system and has been used primarily to prevent rejection in patients who have had organ transplants. Daclizumab has fewer side effects than other immune suppressant drugs.

Patients with ITP 18 years of age or older who have platelet counts less than 30,000/microliter and have not responded to prednisone treatment may be eligible for this study. Candidates will be screened with a medical history, physical examination, and blood tests.

Participants will have a 15-minute infusion of daclizumab every 2 weeks for five doses. They will be seen by a physician at least once every 2 weeks while receiving the drug and then at weeks 12, 20, and 32 of the study. Blood will be drawn at the 4- and 8-week visits during treatment for diagnostic tests, and at each follow-up visit after treatment to assess the response to therapy.

Patients who respond well to treatment will have their pre-study immunosuppressive medicines tapered gradually one at a time starting with the 1-month follow-up visit. If their platelet count falls to pre-treatment levels at any time during the tapering, the dose reduction will stop and pre-study medications will be re-started, if necessary.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an acquired blood disease in which the individual's immune system destroys platelets, the blood cells responsible for clotting. A number of standard treatments exist to decrease the destruction of platelets, including drugs such as the steroid hormone prednisone, or removal of the spleen. Over a third of adult patients will not maintain adequate platelet counts with these treatments. Alternative treatments may be indicated due to bleeding symptoms or baseline platelet counts less than 20,000/ul, a level at which spontaneous serious bleeding can occur. Therapy for chronic ITP is generally effective in less than 30-50% of patients, however, and most of these agents have significant toxicities with long-term use, are expensive, or their administration interferes with daily activities.

Daclizumab is a humanized anti-interleukin-2 receptor monoclonal antibody that works by targeting and impairing activated T lymphocytes, a subset of white blood cells that has been thought to be involved in the development and maintenance of ITP. Daclizumab is a well-tolerated and time-limited therapy, and is easily administered on an outpatient basis. The purpose of this study is to test the efficacy of daclizumab as either a sole agent in the treatment of chronic, symptomatic ITP, or as a treatment that might allow a decrease or discontinuation of medications such as prednisone.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female greater than or equal to 18 years old

Immune thrombocytopenia, and all of the following:

at least three months since initial diagnosis

lack of sustained response to initial treatment with prednisone, characterized by failure to maintain a platelet count of at least 30,000/ul for at least six weeks using prednisone at a dose of at least 10 mg per day

baseline platelet count (as determined by an average of platelet count values over two months immediately prior to study entry) of less than 30,000/ul

*Note: In patients receiving IVIG or anti-D, platelet values immediately prior to infusion of the drug (i.e., at platelet nadir) will be considered in the determination of the baseline platelet value.

Splenectomy or prior use of second-line immunomodulatory treatments (such as, but not limited to, CSA, danazol, azathioprine or cyclophosphamide) will not be considered a requirement for inclusion.

EXCLUSION CRITERIA:

ECOG performance status greater than 1

Concurrent symptomatic autoimmune hemolysis (Evans syndrome) characterized by hemoglobin less than 10 gm/dl or requirement for more than two units red cells within three months of enrollment, due to hemolysis

Concurrent autoimmune disorders requiring treatment for involvement of organ systems other than cytopenias

Initiation of any new immunomodulator agent, or increase in dose or frequency of any existing immunomodulator agent (such as, but not limited to, CSA, danazol, azathioprine or cyclophosphamide; IVIG and anti-D excepted) within two months of study entry

Autologous transplantation for immune thrombocytopenia within one year of study entry

Concurrent bleeding diathesis

Echinacea use within three months of study entry

Pregnancy or lactation

Chronic or current clinically significant infection, including HIV positivity and acute or persistent hepatitis B and C virus infection (characterized by elevated transaminases and positive hepatitis B surface antigen [HBsAg], or anti-hepatitis C virus [anti-HCV] antibody)

History of active M. Tuberculosis infection

Diagnosis of malignancy (with the exception of non-melanoma skin cancer and other malignancies which by virtue of surgical resection and no recurrence for at least five years prior to enrollment are considered to be cured)

Inadequate mental capacity to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 2002-11; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Berchtold P, Wenger M. Autoantibodies against platelet glycoproteins in autoimmune thrombocytopenic purpura: their clinical significance and response to treatment. Blood. 1993 Mar 1;81(5):1246-50. PMID 8443385
- [Background] He R, Reid DM, Jones CE, Shulman NR. Spectrum of Ig classes, specificities, and titers of serum antiglycoproteins in chronic idiopathic thrombocytopenic purpura. Blood. 1994 Feb 15;83(4):1024-32. PMID 8111044
- [Background] Kiefel V, Freitag E, Kroll H, Santoso S, Mueller-Eckhardt C. Platelet autoantibodies (IgG, IgM, IgA) against glycoproteins IIb/IIIa and Ib/IX in patients with thrombocytopenia. Ann Hematol. 1996 Apr;72(4):280-5. doi: 10.1007/s002770050173. PMID 8624385